CLINICAL TRIAL: NCT04783363
Title: Study Comparing Satisfaction of Hospitalized Patients Receiving Invasive Care for Cancer Treatment, With Snoezelen Session Versus Standard Care (SNOEZELEN)
Brief Title: Study Comparing Satisfaction of Hospitalized Patients Receiving Invasive Care for Cancer Treatment, With Snoezelen Session Versus Standard Care
Acronym: SNOEZELEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-012
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: Supportive care; Snoezelen
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): * Visit 1: with Snoezelen session before invasive care
  * Visit 2: standard care (=without Snoezelen session) before invasive care
  Interventions: Other: Snoezelen session
- Arm B (Experimental): * Visit 1: standard care (=without Snoezelen session) before invasive care
  * Visit 2: with Snoezelen session before invasive care
  Interventions: Other: Snoezelen session

INTERVENTIONS:
Other: Snoezelen session — before one of two repeated invasive care

SUMMARY:
This is a monocentric, comparative, open-label, randomized, crossover study enrolling patients hospitalized in Strasbourg Europe Cancerology Institute, receiving repeated invasive care for cancer treatment.

The purpose of this study is to compare the satisfaction of patients, regarding their perception of care, with or without Snoezelen session.

DETAILED DESCRIPTION:
Patients will followed during two visits for a repeated invasive care. They will be randomized to two groups in a 1:1 ratio.

Crossover plan and arms are described as follow:

Arm A : Visit 1 with Snoezelen session before invasive care and Visit 2 without Snoezelen session before invasive care (standard care)

Arm B : Visit 1 without Snoezelen session before invasive care (standard care) and Visit 2 with Snoezelen session before invasive care

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for cancer and hospitalized for invasive care
* Two programmed hospitalization for repeated care
* Patients receiving one of the following invasive care: Huber needle application (transfusion, parenteral nutrition), complex wound dressing, intrathecal chemotherapy, ascites fluid or pleural puncture
* Patients must be ≥ 18 years old
* Performance Status ≤ 3
* Absence of psychiatric disorder impairing follow-up
* Ability to speak, understand, write and read French
* Signed informed consent from the patient
* Affiliation to social security system

Exclusion Criteria:

* Patients presenting infectious symptoms requiring isolation
* Patients < 18 years old or patients ≥ 18 years old under supervision
* Patients placed under judicial protection or guardianship
* Women that are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction regarding their perception of care quality (with or without Snoezelen session) at Visit 1 | immediately after invasive care at Visit 1
  Evaluation using a modified Visual Analog Scales, Oberts, 1984
Patient satisfaction regarding their perception of care quality (with or without Snoezelen session) at Visit 2 | immediately after invasive care at Visit 2
  Evaluation using a modified Visual Analog Scales, Oberts, 1984

SECONDARY OUTCOMES:
Change in patient perceived pain, with or without Snoezelen session | At admission (i.e. before Snoezelen session, if applicable) and immediately after invasive care at Visit n°1; At admission (i.e. before Snoezelen session, if applicable) and immediately after invasive care at Visit n°2
  Numeric visual analog scale (0 to 10)
Change in patient perceived anxiety, with or without Snoezelen session | At admission (i.e. before Snoezelen session, if applicable) and immediately after invasive care at Visit n°1; At admission (i.e. before Snoezelen session, if applicable) and immediately after invasive care at Visit n°2
  Numeric visual analog scale (0 to 10)
Comparing relationship between patient and caregiver, with or without Snoezelen session | immediately after invasive care at Visit 1 ; immediately after invasive care at Visit 2
  Numeric visual analog scale (0 to 10)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France